CLINICAL TRIAL: NCT04904952
Title: Effect of N-acetylcysteine as Add on Therapy With Selective Serotonin Reuptake Inhibitors in Moderate to Severe Obsessive Compulsive Disorder Patients
Brief Title: Effect of N-acetylcysteine as Add on Therapy With SSRI in Moderate to Severe OCD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Sadia Binte Anwar Sonia, MD, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU/2021/2300
Record Dates: First submitted 2021-05-23; First posted 2021-05-27 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: OCD
Keywords: N-acetylcysteine, OCD, MRS, Glutamate
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): This arm includes 30 OCD patients receiving SSRIs
  Interventions: Drug: N-acetylcysteine tablet 600mg
- Control (Placebo Comparator): This arm includes 30 OCD patients receiving SSRIs
  Interventions: Drug: Placebo tablet 600mg

INTERVENTIONS:
Drug: N-acetylcysteine tablet 600mg — N-acetylcysteine tablet 600mg/day and doubling weekly to reach a maximum dose of 2400mg/day (at week-3) for remaining 7 weeks along with SSRIs
  Arms: Experimental
Drug: Placebo tablet 600mg — Placebo tablet 600mg/day and doubling weekly to reach a maximum dose of 2400mg/day (at week-3) for remaining 7 weeks along with SSRIs
  Arms: Control

SUMMARY:
Title:

Effect of n-acetylcysteine as add-on therapy with Selective Serotonin Reuptake Inhibitors in moderate to severe Obsessive Compulsive Disorder patients.

Purpose of the study:

To assess the effects of the addition of n-acetylcysteine with SSRIs on the severity of symptoms in obsessive-compulsive disorder patients.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is the fourth most common mental disorder in Bangladesh and around the world. Selective serotonin reuptake inhibitors (SSRIs) are commonly administered drugs for treating children and adolescents with OCD. The treatment of this condition has remained unsatisfactory, only 40-60% of patients with OCD respond to SSRIs, and about 40 to 60% of patients with OCD do not completely respond to this drug. Researchers throughout the world are involved to obtain new pharmacotherapy for the treatment of OCD. A good number of evidences have proved that glutamate plays a significant role in the pathophysiology of OCD.N-acetylcysteine (NAC) is an amino acid derivative, is a health supplement, and has neuroprotective effects that target the glutamatergic system. Some recent trials attempted to assess the effect of n-acetylcysteine as an add-on therapy with SSRIs to improve symptoms in OCD patients. Aim: This proposed study is therefore an effort whether there is any role of n-acetylcysteine adjuncts with SSRI produce better improvement than SSRI alone in OCD patients. Method: This study will be a randomized, double-blind, placebo-controlled multicenter trial that will be conducted in the department of pharmacology, BSMMU in collaboration with the department of psychiatry, BSMMU, and Combined Military Hospital (CMH), Dhaka from the day of approval by the IRB to January 2022. A total of 56 patients suffering from OCD will be selected according to inclusion and exclusion criteria. The diagnosis of patients suffering from OCD and the selection of drug and dosage would be performed by a senior professor of the psychiatry department. After completing the necessary formalities including informed consent of the patients, the patient would undergo a selected questionnaire Yale-Brown Obsessive Scale (Y-BOCS-10) to assess the severity of the disease. The patients would be randomly allocated into two arms: control and intervention. Patients in the intervention arm would consist of 30 patients who will receive SSRIs plus NAC. NAC was titrated from 600mg/day and doubling weekly to reach a maximum dose of 2400mg/day (at week-3) for the remaining 7 weeks. On the other hand, the control arm would consist of 30 patients who will receive SSRIs plus a placebo for 10 weeks. The severity of symptoms will be assessed after 4 weeks and 10 weeks follow-up. The brain glutamate level, ALT, AST, serum creatinine, and ECG will be measured at baseline and after 10 weeks. The regularity of medicine intake will be ensured over the telephone, pill count, and from the patient's compliance sheet. Statistical analysis will be obtained by SPSS (statistical package for social science) version 24. Paire't' test will be done to compare between two means of before and after the intervention. Proportion test 'Z' will be done to compare the proportion between the intervention group and the placebo group. The calculated 'p' value may suggest the level of significance (significant at p<0.05). Ethical consideration: After approval from IRB every eligible patient will be informed about the intervention and the study objectives. Patients will also be informed that they can participate or to withdraw at any time without compromising their medical care. Patient confidentiality will be strictly maintained. Patient's personal data regarding the name, age, sex, and other information will not be disclosed anywhere and will be used only for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed OCD patients diagnosed by Psychiatric Consultant of the Department of Psychiatry according to DSM-5 criteria (Appendix VI).
* Moderate to severe OCD patients having AY-BOCS score > 16
* Age: 18 years or above
* Sex: Both male and female

Exclusion Criteria:

Patients receiving antidepressant within last two months.

* Patients having any history of psychiatric and medical conditions will be excluded from the study.
* Patients having suicidal thoughts.
* Pregnancy and lactation.
* Patients who are receiving psychotherapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2022-01-10 (Estimated); Study Completion 2022-01-10 (Estimated)

PRIMARY OUTCOMES:
OCD severity score assessment | 10 weeks
  Assess the severity score of OCD symptoms by YBOCS-10 at baseline, after 4 weeks, and after10 weeks.
  And compare the score between two groups. YBOCS-10 range from 0-40 with the following scores: 0-14 Non significant to mild, 15-23 Mild to moderate, 23-29 Moderate to severe, 30-40 Severe to disabling.

SECONDARY OUTCOMES:
Neurochemical assessment | 10 weeks
  To estimate the brain glutamate level by Magnetic Resonance Spectroscopy (MRS) at baseline and after 10 weeks supplementation of n-acetylcysteine and SSRI. To compare the brain glutamate level by Magnetic Resonance Spectroscopy (MRS) at baseline and after 10 weeks supplementation of n-acetylcysteine and SSRI.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Md. Sayedur Rahman, MBBS, M.Phil, Study Chair — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (2):
- Bangladesh (2):
  - BSMMU, Dhaka
  - Sadia Binte Anwar Sonia, Dhaka